CLINICAL TRIAL: NCT00075218
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study Of SU011248 In The Treatment Of Patients With Imatinib Mesylate (Gleevec Tm, Glivec)-Resistant Or Intolerant Malignant Gastrointestinal Stromal Tumor
Brief Title: A Study To Assess The Safety And Efficacy Of SU11248 In Patients With Gastrointestinal Stromal Tumor(GIST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A6181004; NCT00085618 (obsolete NCT alias)
Record Dates: First submitted 2004-01-06; First posted 2004-01-08 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-08

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Placebo Comparator)
  Interventions: Drug: Placebo
- A (Active Comparator)
  Interventions: Drug: SU011248

INTERVENTIONS:
Drug: Placebo — 50 mg taken orally once a day. 6 week treatment cycle (Schedule 4/2) 4 weeks on study drug/2 weeks off study drug.
  Arms: B
Drug: SU011248 — 50 mg taken orally once a day. 6 week treatment cycle (Schedule 4/2) 4 weeks on study drug/2 weeks off study drug.
  Arms: A

SUMMARY:
A study to assess the safety and efficacy of SU11248 in patients with gastrointestinal stromal tumor (GIST) whose disease has failed imatinib therapy or who were intolerant to imatinib treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically-proven diagnosis of malignant GIST not amenable to surgery, radiation or combined modality treatment with curative intent
* Failed Gleevec treatment or intolerant to Gleevec therapy

Key Exclusion Criteria:

* Treatment with any chemotherapy, chemoembolization therapy, immunotherapy, or investigational agent since the last dose of Gleevec

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2003-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (53):
- United States (23):
  - Pfizer Investigational Site, Duarte, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Columubs, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
- Australia (7):
  - Pfizer Investigational Site, Garran, Australian Capital Territory
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, Auchenflower, Queensland
  - Pfizer Investigational Site, Ashford, South Australia
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, East Melbourne, Victoria
- Pfizer Investigational Site, Leuven, Belgium
- Canada (2):
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- France (3):
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Villejuif
- Italy (6):
  - Pfizer Investigational Site, Aviano, PN
  - Pfizer Investigational Site, Candiolo, Torino
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Torino
- Netherlands (2):
  - Pfizer Investigational Site, Groningen, Provincie Groningen
  - Pfizer Investigational Site, Rotterdam, South Holland
- Pfizer Investigational Site, Singapore, Singapore
- Spain (3):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet Del Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
- Pfizer Investigational Site, Lausanne, Switzerland
- United Kingdom (4):
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Demetri GD, van Oosterom AT, Garrett CR, Blackstein ME, Shah MH, Verweij J, McArthur G, Judson IR, Heinrich MC, Morgan JA, Desai J, Fletcher CD, George S, Bello CL, Huang X, Baum CM, Casali PG. Efficacy and safety of sunitinib in patients with advanced gastrointestinal stromal tumour after failure of imatinib: a randomised controlled trial. Lancet. 2006 Oct 14;368(9544):1329-38. doi: 10.1016/S0140-6736(06)69446-4. PMID 17046465
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181004&StudyName=A%20Study%20To%20Assess%20The%20Safety%20And%20Efficacy%20Of%20SU11248%20In%20Patients%20With%20Gastrointestinal%20Stromal%20Tumors%20%28GIST%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began (medical clinic) in December 2003. Study was unblinded on 27 January 2005 (end of Double-blind treatment). Subjects experiencing disease progression could crossover to Open-label treatment. Open-label data collection ended May 2008.
Pre-assignment Details: 361 subjects randomized to double-blind treatment in 2:1 ratio (sunitinib vs. Placebo).
  255 subjects continued on or crossed over to Open-label treatment.
Groups:
- Sunitinib Double-Blind Treatment: Starting dose: 50 mg orally once daily as a single agent for 4 consecutive weeks followed by a 2-week off-treatment period to form a complete cycle of 6 weeks. (Schedule 4/2). Subjects received best supportive care in addition to the study treatment.
- Placebo Double-Blind Treatment: Starting daily dose of 1 capsule, size- and color-matched to the sunitinib 50-mg capsule for 4 consecutive weeks followed by a 2-week off-treatment period to form a complete cycle of 6 weeks (Schedule 4/2). Subjects received best supportive care in addition to the study treatment. Subjects were provided the opportunity to receive open-label sunitinib at the time of confirmed disease progression or study unblinding.
- Sunitinib Open-Label Treatment: Subjects experiencing disease progression could have their treatment assignment unblinded, and subjects who had been receiving placebo could crossover to open-label treatment with sunitinib; subjects who had been receiving sunitinib during double-blind treatment of the study could continue to do so after unblinding if, in the opinion of the investigator, there was sufficient evidence of clinical benefit.
Period: Double-Blind Treatment
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment | Sunitinib Open-Label Treatment
Started | 243 (Intent To Treat Population (ITT)) | 118 (Intent To Treat Population (ITT)) | 0
Received Double-Blind Treatment | 228 (As Treated Population (AT)) | 114 (As Treated Population (AT)) | 0
Crossed Over to Open-Label Treatment | 152 | 103 | 0
Completed | 152 (Defined:subjects completed double-blind treatment phase and/or entered open-label treatment phase.) | 103 (Defined:subjects completed double-blind treatment phase and/or entered open-label treatment phase.) | 0
Not Completed | 91 | 15 | 0
Not completed — Adverse Event | 23 | 4 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 58 | 6 | 0
Not completed — Decision of Sponsor | 0 | 1 | 0
Not completed — No study medication taken | 2 | 0 | 0
Period: Open-Label Treatment
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment | Sunitinib Open-Label Treatment
Started | 0 | 0 | 255
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 255
Not completed — Lack of Efficacy | 0 | 0 | 174
Not completed — Adverse Event | 0 | 0 | 51
Not completed — Withdrawal by Subject | 0 | 0 | 12
Not completed — Decision of Sponsor | 0 | 0 | 8
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — enrolled in a separate continuation | 0 | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment | Total
Number analyzed (Participants) | 243 | 118 | 361
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 170 | 81 | 251.0
  >=65 years | 73 | 37 | 110.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 71 | 162.0
  Male | 152 | 47 | 199.0

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression (TTP) as Assessed by Imaging Studies at End of Double-blind Treatment Phase
Description: Time from randomization to first documentation of objective tumor progression based on the assessment of an independent, third-party imaging laboratory using RECIST (Response Evaluation Criteria in Solid Tumors).
Time Frame: Day 28 of each 6-week cycle : duration of double-blind treatment phase
Population: From the Intent to Treat (ITT) population, 82 subjects on sunitinib treatment were observed to have disease progression during blinded phase and were included in TTP analysis. 67 subjects on placebo were observed to have disease progression during blinded phase.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 207 | 105
weeks | 27.3 [16.0 to 32.1] | 6.4 [4.4 to 10]
Statistical Analysis 1: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; The study was designed to test the null hypothesis that the median TTP from placebo treatment is 4 months versus the alternative hypothesis that the median TTP from sunitinib treatment is at least 6 months with an overall 2-sided significance level of 0.05 and power of 90%; Test type: Superiority or Other; p < 0.001, Log Rank — The nominal levels of significance for the interim and final analyses were determined at the time of the analyses using the Lan-DeMets procedure with an O'Brien-Fleming stopping rule; two-sided unstratified log-rank test; Hazard Ratio (HR) = 0.329, 95% CI [0.233 to 0.466]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time from randomization to first documentation of objective tumor progression or to death due to any cause (on treatment or within 28 days of last dose).
Time Frame: Day 28 of each cycle : duration of double-blind treatment phase
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
weeks | 22.9 [10.9 to 28.0] | 6.0 [4.4 to 9.7]
Statistical Analysis 1: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; Test type: Superiority or Other; p < 0.001, Log Rank — No p-value adjustment for multiple comparisons; Hazard Ratio (HR) = 0.347, 95% CI [0.253 to 0.475]

3. Secondary Outcome: Overall Survival Status of Subjects
Description: Number of subjects alive at end of study.
Time Frame: clinic visit or telephone contact every 2 months for up to 3 years from the last dose of study drug
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
participants
  Dead | 176 | 90
  Alive | 67 | 28

4. Secondary Outcome: Overall Survival
Description: Time from date of randomization to date of death due to any cause.
Time Frame: clinic visit or telephone contact every 2 months for up to 3 years from the last dose of study drug
Population: ITT population; Number subjects Dead = 176, 90 (sunitinib, placebo respectively). Subjects who were not known to be dead at the time the database was closed for analysis were censored on the date they were last known to be alive.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
weeks | 72.7 [61.3 to 83.0] | 64.9 [45.7 to 96.0]
Statistical Analysis 1: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; Test type: Superiority or Other; p = 0.306, Log Rank — No p-value adjustment for multiple comparisons; Hazard Ratio (HR) = 0.876, 95% CI [0.679 to 1.129]

5. Secondary Outcome: Overall Survival Based on the Rank Preserving Structural Failure Time Method
Description: time from date of randomization to date of death due to any cause (rank preserving structural failure time method).
Time Frame: clinic visit or telephone contact every 2 months for up to 3 years from the last dose of study drug
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
weeks | 72.7 [61.3 to 83.0] | 39.0 [28.0 to 54.1]
Statistical Analysis 1: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; Test type: Superiority or Other; p = 0.306, Rank Preserving Structural Failure Time — No p-value adjustment for multiple comparisons; Hazard Ratio (HR) = 0.505, 95% CI [0.262 to 1.134] — 95% CI for Hazard Ratio is from 2.5% and 97.5% Empirical Percentiles of 100,000 Bootstraps

6. Secondary Outcome: Best Overall Tumor Response During Double-blind Treatment Phase
Description: Tumor response according to Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Day 28 of each cycle : duration of double-blind treatment phase
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 16 | 0
  Stable Disease | 128 | 50
  Progressive Disease | 45 | 44
  Unable to Evaluate | 1 | 0
  Missing | 53 | 24

7. Secondary Outcome: Confirmed Objective Response (CR or PR) in Subjects
Description: Overall confirmed objective response = confirmed Complete Response (CR) OR confirmed Partial Response (PR) according to RECIST. Confirmed responses were those that persisted on repeat imaging study ≥ 4 weeks after initial documentation of response.
Time Frame: Day 28 of each cycle : duration of double-blind treatment phase
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
participants | 16 | 0
Statistical Analysis 1: Comparison: Sunitinib Double-Blind Treatment; Test type: Superiority or Other; rate (percentage) = 6.6, 95% CI [3.8 to 10.5] — Used exact method based on binomial distribution
Statistical Analysis 2: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; Test type: Superiority or Other; p = 0.004, Pearson chi-square test — No p-value adjustment for multiple comparisons; Treatment Difference (%) = 6.58, 95% CI [3.47 to 9.70]

8. Secondary Outcome: Time to Tumor Response (TTR)
Description: Time from date of randomization to first documentation of objective tumor response that was subsequently confirmed. TTR was only calculated for the subgroup of subjects with a confirmed objective tumor response.
Time Frame: Day 28 of each cycle : duration of double-blind treatment phase
Population: ITT population. Number of subjects analyzed = number of subjects with tumor response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 16 | 0
weeks | 13.4 [9.9 to 16.1] |

9. Secondary Outcome: Duration of Performance Status Maintenance
Description: Time from randomization until the last time the performance status was no worse than at baseline or to death due to cancer in the absence of previous documentation of performance status worsening.
Time Frame: Day 28 of each cycle : duration of double-blind treatment phase
Population: ITT Population. Number of subjects at median observed to have status worsening or died before status worsening.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 106 | 0
weeks | 18.9 [12.1 to 31.1] |

10. Primary Outcome: Time to Tumor Progression (TTP) as Assessed in the Double-blind Treatment Phase at End of Study
Description: as for outcome 1
Time Frame: Day 28 of each 6-week cycle : duration of double-blind treatment phase after Last Subject Last Visit (LSLV)
Population: From the Intent to Treat (ITT) population, 91 subjects on sunitinib treatment were observed to have disease progression during blinded phase and were included in TTP analysis. 73 subjects on placebo were observed to have disease progression during blinded phase.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
weeks | 26.6 [16.0 to 32.1] | 6.4 [4.4 to 10.0]
Statistical Analysis 1: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; Test type: Superiority or Other; p < 0.001, Log Rank — two-sided unstratified log-rank test; Hazard Ratio (HR) = 0.339, 95% CI [0.244 to 0.472]
Statistical Analysis 2: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; Stratified log-rank test; Test type: Superiority or Other; p < 0.001, Log Rank; log-rank test of treatment stratified by prior imatinib mesylate response and McGill Pain Questionnaire's Present Pain Intensity score; Hazard Ratio (HR) = 0.327, 95% CI [0.232 to 0.460]

11. Secondary Outcome: Time to Pain Progression Using McGill Pain Questionnaire-present Pain Intensity (MPQ-PPI)
Description: 25th Quartile: Time to Progression. Progression: a) No change (NC) in MPQ-PPI score (0=no pain to 5=excruciating pain) with increase total analgesic use >= 50% over baseline OR b) Increase score >= 1 point with either NC in total analgesic use or increase total analgesic use >= 50% over baseline. (50th Quartile not achieved.)
Time Frame: Day 1 & 28 of each cycle : duration of double-blind treatment phase
Population: Pain-Relief-Response population. Subjects at 25th Quartile with pain progress during blinded phase.
Measure: Median (95% Confidence Interval); unit: weeks (25th Quartile)
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 37 | 0
weeks (25th Quartile) | 12.1 [6.1 to 27.1] |
Statistical Analysis 1: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; Test type: Superiority or Other; p = 0.9322, Log Rank; 2-sided, unstratified log-rank test; Hazard Ratio (HR) = 0.972, 95% CI [0.508 to 1.860]

12. Secondary Outcome: Subjects With Pain Relief Response Using McGill Pain Questionnaire-present Pain Intensity (MPQ-PPI)
Description: MPQ-PPI: 0=no pain to 5= excruciating pain. Pain Relief Response= 1) Decrease by >= 1 points in MPQ-PPI score with either Decrease or No Change in total analgesic use >= 50% over baseline OR 2) No change in MPQ-PPI score with Decrease total analgesic use >= 50% over baseline.
Time Frame: Day 1 & 28 of each cycle : duration of double-blind treatment phase
Population: Pain-Relief-Response population.
Measure: Number; unit: participants
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 150 | 75
participants | 46 | 10
Statistical Analysis 1: Comparison: Sunitinib Double-Blind Treatment vs Placebo Double-Blind Treatment; Test type: Superiority or Other; p = 0.0046, Pearson chi-square; Treatment Difference (percent) = 17.3, 95% CI [6.7 to 28.0] — 95% CI of Difference based on normal distribution. Percent = (number of subjects with response per total subjects per treatment in defined analysis population)*100

13. Secondary Outcome: Change From Baseline Score in EuroQoL Visual Analog Scale (EQ-VAS)
Description: Change: median score at observation minus median score at baseline. EQ-VAS score on the self-rated "thermometer," indicating the patient's own assessment of their health status from 0 (worst) to 100 (best) imaginable health state.
Time Frame: Day 1 & 28 of each cycle : duration of double-blind treatment phase
Population: ITT population. Number subjects with evaluable data: (n=sunitinib, placebo)
Measure: Median (Full Range); unit: score on scale
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
score on scale
  Cycle 1 Day 28 (n=187, 89) | -3.0 [-60.0 to 70.0] | 0.0 [-50.0 to 45.0]
  Cycle 2 Day 1 (n=148, 53) | 0.0 [-60.0 to 55.0] | 0.0 [-30.0 to 41.0]
  Cycle 2 Day 28 (n=132, 41) | -4.5 [-50.0 to 55.0] | 0.0 [-80.0 to 40.0]
  Cycle 3 Day 1 (n=102,16) | 0.0 [-58.0 to 32.0] | 0.0 [-75.0 to 34.0]
  Cycle 3 Day 28 (n=91,13) | -5.0 [-55.0 to 42.0] | -1.0 [-75.0 to 16.0]
  Cycle 4 Day 1 (n=73,10) | 0.0 [-65.0 to 40.0] | 5.0 [-10.0 to 15.0]

14. Secondary Outcome: Change From Baseline in EQ-5D Health State Profile Index
Description: Change: median index score at observation minus median index score at baseline. EQ-5D is a generic instrument that describes health status in 5 dimensions (mobility, self-care, pain/discomfort, anxiety/depression, usual activities) with a weighted health Index based on general population values where where 0.0 = death and 1.0 = perfect health.
Time Frame: Day 1 & 28 of each cycle : duration of double-blind treatment phase
Population: ITT Population. Number subjects with evaluable data: (n=sunitinib, placebo)
Measure: Median (Full Range); unit: score on scale
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment
Number analyzed (Participants) | 243 | 118
score on scale
  Cycle 1 Day 28 (n=185, 87) | 0.000 [-1.008 to 0.736] | 0.000 [-0.655 to 0.532]
  Cycle 2 Day 1 (n=149, 53) | 0.000 [-1.244 to 0.603] | 0.000 [-0.603 to 0.434]
  Cycle 2 Day 28 (n=129, 41) | -0.017 [-1.008 to 0.603] | 0.000 [-0.694 to 0.655]
  Cycle 3 Day 1 (n=104, 17) | 0.000 [-0.694 to 0.639] | 0.000 [-0.655 to 0.192]
  Cycle 3 Day 28 (n=91, 13) | -0.036 [-1.175 to 0.736] | 0.000 [-0.655 to 0.204]
  Cycle 4 Day 1 (n=74, 10) | 0.000 [-0.768 to 0.603] | 0.059 [-0.152 to 0.275]

ADVERSE EVENTS:
Arm/Group | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment | Sunitinib Open-Label Treatment
Serious Adverse Events (participants affected / at risk) | 83 | 27 | 122
Other Adverse Events (participants affected / at risk) | 223 | 110 | 254
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment | Sunitinib Open-Label Treatment
Anaemia (Blood and lymphatic system disorders) | 11/228 | 1/114 | 10/255
Thrombocytopenia (Blood and lymphatic system disorders) | 5/228 | 0/114 | 4/255
Neutropenia (Blood and lymphatic system disorders) | 2/228 | 0/114 | 1/255
Febrile neutropenia (Blood and lymphatic system disorders) | 1/228 | 0/114 | 1/255
Leukopenia (Blood and lymphatic system disorders) | 1/228 | 0/114 | 1/255
Cardiac arrest (Cardiac disorders) | 1/228 | 1/114 | 0/255
Cardiac disorder (Cardiac disorders) | 1/228 | 0/114 | 0/255
Cardiac failure (Cardiac disorders) | 1/228 | 1/114 | 0/255
Cardiomyopathy (Cardiac disorders) | 1/228 | 0/114 | 0/255
Ejection fraction decreased (Cardiac disorders) | 1/228 | 0/114 | 0/255
Left ventricular failure (Cardiac disorders) | 1/228 | 0/114 | 0/255
Mitral valve imcompetence (Cardiac disorders) | 1/228 | 0/114 | 0/255
Pyloric stenosis (Congenital, familial and genetic disorders) | 1/228 | 0/114 | 0/255
Hypothyroidism (Endocrine disorders) | 1/228 | 0/114 | 4/255
Abdominal pain (Gastrointestinal disorders) | 13/228 | 6/114 | 29/255
Nausea (Gastrointestinal disorders) | 5/228 | 3/114 | 8/255
Vomiting (Gastrointestinal disorders) | 5/228 | 4/114 | 12/255
Ascites (Gastrointestinal disorders) | 4/228 | 1/114 | 3/255
Diarrhoea (Gastrointestinal disorders) | 4/228 | 0/114 | 4/255
Abdominal distension (Gastrointestinal disorders) | 2/228 | 0/114 | 3/255
Constipation (Gastrointestinal disorders) | 2/228 | 1/114 | 5/255
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2/228 | 3/114 | 4/255
Intestinal obstruction (Gastrointestinal disorders) | 2/228 | 1/114 | 2/255
Melaena (Gastrointestinal disorders) | 2/228 | 0/114 | 1/255
Abdominal pain upper (Gastrointestinal disorders) | 1/228 | 0/114 | 1/255
Anal fistula (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Gastric haemorrhage (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Gastric ulcer (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Gastritis (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Gastritis haemorrhagic (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Gastrointestinal obstruction (Gastrointestinal disorders) | 1/228 | 1/114 | 0/255
Haematemesis (Gastrointestinal disorders) | 1/228 | 1/114 | 3/255
Haemorrhoids (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Intestinal haemorrhage (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Oesophageal haemorrhage (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Rectal haemorrhage (Gastrointestinal disorders) | 1/228 | 1/114 | 5/255
Small intestinal obstruction (Gastrointestinal disorders) | 1/228 | 0/114 | 3/255
Ileus (Gastrointestinal disorders) | 0/228 | 2/114 | 2/255
Subileus (Gastrointestinal disorders) | 0/228 | 1/114 | 1/255
Disease progression (General disorders) | 8/228 | 4/114 | 33/255
Pyrexia (General disorders) | 8/228 | 1/114 | 11/255
Fatigue (General disorders) | 2/228 | 1/114 | 3/255
Oedema peripheral (General disorders) | 2/228 | 0/114 | 0/255
Asthenia (General disorders) | 1/228 | 1/114 | 3/255
Chills (General disorders) | 1/228 | 0/114 | 2/255
Drug interaction (General disorders) | 1/228 | 0/114 | 0/255
General physical health deterioration (General disorders) | 1/228 | 3/114 | 4/255
Multi-organ failure (General disorders) | 1/228 | 0/114 | 1/255
Oedema (General disorders) | 1/228 | 0/114 | 0/255
Chest pain (General disorders) | 0/228 | 1/114 | 3/255
Acute hepatic failure (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Bile duct stone (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Cholecystitis acute (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Cholelithiasis (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Cholestasis (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Hepatic failure (Hepatobiliary disorders) | 1/228 | 0/114 | 2/255
Hepatic function abnormal (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Hepatic haemorrhage (Hepatobiliary disorders) | 1/228 | 0/114 | 1/255
Catheter sepsis (Infections and infestations) | 1/228 | 0/114 | 0/255
Central line infection (Infections and infestations) | 1/228 | 0/114 | 0/255
Infection (Infections and infestations) | 1/228 | 0/114 | 3/255
Mediastinitis (Infections and infestations) | 1/228 | 0/114 | 0/255
Pneumonia (Infections and infestations) | 1/228 | 1/114 | 4/255
Staphylococcal sepsis (Infections and infestations) | 1/228 | 0/114 | 0/255
Urinary tract infection (Infections and infestations) | 1/228 | 0/114 | 2/255
Viral infection (Infections and infestations) | 1/228 | 1/114 | 0/255
Bacteraemia (Infections and infestations) | 0/228 | 1/114 | 2/255
Cystitis (Infections and infestations) | 0/228 | 1/114 | 0/255
Lower respiratory tract infection (Infections and infestations) | 0/228 | 1/114 | 1/255
Wound dehiscence (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 0/255
Aspartate aminotransferase increased (Investigations) | 1/228 | 0/114 | 0/255
Blood creatinine increased (Investigations) | 1/228 | 0/114 | 3/255
Haemoglobin decreased (Investigations) | 1/228 | 1/114 | 2/255
Dehydration (Metabolism and nutrition disorders) | 4/228 | 0/114 | 10/255
Hypoglycaemia (Metabolism and nutrition disorders) | 4/228 | 0/114 | 0/255
Food intolerance (Metabolism and nutrition disorders) | 1/228 | 0/114 | 0/255
Hypercalcaemia (Metabolism and nutrition disorders) | 1/228 | 1/114 | 1/255
Hypocalcaemia (Metabolism and nutrition disorders) | 1/228 | 0/114 | 1/255
Hypokalaemia (Metabolism and nutrition disorders) | 1/228 | 0/114 | 1/255
Anorexia (Metabolism and nutrition disorders) | 0/228 | 1/114 | 3/255
Appetite disorder (Metabolism and nutrition disorders) | 0/228 | 1/114 | 0/255
Back pain (Musculoskeletal and connective tissue disorders) | 1/228 | 2/114 | 1/255
Fistula (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 0/255
Flank pain (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 0/255
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 0/255
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 1/255
Bone pain (Musculoskeletal and connective tissue disorders) | 0/228 | 1/114 | 0/255
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/228 | 1/114 | 0/255
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0/228 | 1/114 | 0/255
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/228 | 0/114 | 3/255
Haemorrhagic tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 1/114 | 0/255
Cerebral ischaemia (Nervous system disorders) | 1/228 | 0/114 | 0/255
Encephalopathy (Nervous system disorders) | 1/228 | 0/114 | 0/255
Myoclonus (Nervous system disorders) | 1/228 | 0/114 | 0/255
Somnolence (Nervous system disorders) | 1/228 | 0/114 | 2/255
Syncope (Nervous system disorders) | 1/228 | 0/114 | 3/255
Transient ischaemic attack (Nervous system disorders) | 1/228 | 0/114 | 1/255
Cerebrovascular accident (Nervous system disorders) | 0/228 | 1/114 | 1/255
Paralysis (Nervous system disorders) | 0/228 | 1/114 | 0/255
Insomnia (Psychiatric disorders) | 0/228 | 1/114 | 0/255
Nervousness (Psychiatric disorders) | 0/228 | 1/114 | 0/255
Haematuria (Renal and urinary disorders) | 1/228 | 0/114 | 0/255
Nephrotic syndrome (Renal and urinary disorders) | 1/228 | 0/114 | 0/255
Oliguria (Renal and urinary disorders) | 1/228 | 0/114 | 1/255
Renal colic (Renal and urinary disorders) | 1/228 | 0/114 | 0/255
Renal failure acute (Renal and urinary disorders) | 1/228 | 1/114 | 1/255
Urinary retention (Renal and urinary disorders) | 1/228 | 0/114 | 2/255
Hydronephrosis (Renal and urinary disorders) | 0/228 | 1/114 | 0/255
Pelvic pain (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4/228 | 1/114 | 2/255
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Rash (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 0/255
Deep vein thrombosis (Vascular disorders) | 1/228 | 0/114 | 3/255
Haemorrhage (Vascular disorders) | 1/228 | 0/114 | 0/255
Hypertensive crisis (Vascular disorders) | 1/228 | 0/114 | 0/255
Thrombosis (Vascular disorders) | 1/228 | 0/114 | 0/255
Circulatory collapse (Vascular disorders) | 0/228 | 1/114 | 0/255
Haemolytic anaemia (Blood and lymphatic system disorders) | 0/228 | 0/114 | 1/255
Lymphopenia (Blood and lymphatic system disorders) | 0/228 | 0/114 | 1/255
Cardio-respiratory arrest (Cardiac disorders) | 0/228 | 0/114 | 2/255
Angina pectoris (Cardiac disorders) | 0/228 | 0/114 | 1/255
Bradycardia (Cardiac disorders) | 0/228 | 0/114 | 1/255
Cardiac failure congestive (Cardiac disorders) | 0/228 | 0/114 | 1/255
Myocardial infarction (Cardiac disorders) | 0/228 | 0/114 | 1/255
Pericardial effusion (Cardiac disorders) | 0/228 | 0/114 | 1/255
Ventricular hypokinesia (Cardiac disorders) | 0/228 | 0/114 | 1/255
Epidermolysis (Congenital, familial and genetic disorders) | 0/228 | 0/114 | 1/255
Abdominal discomfort (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Anal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Duodenal fistula (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Duodenal ulcer (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Dyspepsia (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Enterocutaneous fistula (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Inguinal hernia (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Large intestinal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Peritoneal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Tongue haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Performance status decreased (General disorders) | 0/228 | 0/114 | 2/255
Catheter related complication (General disorders) | 0/228 | 0/114 | 1/255
Impaired healing (General disorders) | 0/228 | 0/114 | 1/255
Infusion site extravasation (General disorders) | 0/228 | 0/114 | 1/255
Mucosal inflammation (General disorders) | 0/228 | 0/114 | 1/255
Pain (General disorders) | 0/228 | 0/114 | 1/255
Pneumatosis (General disorders) | 0/228 | 0/114 | 1/255
Ulcer haemorrhage (General disorders) | 0/228 | 0/114 | 1/255
Cholecystitis (Hepatobiliary disorders) | 0/228 | 0/114 | 1/255
Hepatotoxicity (Hepatobiliary disorders) | 0/228 | 0/114 | 1/255
Gastroenteritis (Infections and infestations) | 0/228 | 0/114 | 2/255
Abdominal abscess (Infections and infestations) | 0/228 | 0/114 | 1/255
Bacterial infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Campylobacter infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Cellulitis (Infections and infestations) | 0/228 | 0/114 | 1/255
Empyema (Infections and infestations) | 0/228 | 0/114 | 1/255
Gastrointestinal infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Liver abscess (Infections and infestations) | 0/228 | 0/114 | 1/255
Perirectal abscess (Infections and infestations) | 0/228 | 0/114 | 1/255
Respiratory tract infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Sepsis (Infections and infestations) | 0/228 | 0/114 | 1/255
Urosepsis (Infections and infestations) | 0/228 | 0/114 | 1/255
Device malfunction (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Feeding tube complication (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Medication error (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Neck injury (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Skin laceration (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Ammonia increased (Investigations) | 0/228 | 0/114 | 1/255
Blood bilirubin increased (Investigations) | 0/228 | 0/114 | 1/255
Blood creatine phosphokinase increased (Investigations) | 0/228 | 0/114 | 1/255
Blood potassium decreased (Investigations) | 0/228 | 0/114 | 1/255
Blood pressure increased (Investigations) | 0/228 | 0/114 | 1/255
Weight decreased (Investigations) | 0/228 | 0/114 | 1/255
Cachexia (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Hypochloraemia (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Hyponatraemia (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 3/255
Myalgia (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Neck pain (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Hepatic encephalopathy (Nervous system disorders) | 0/228 | 0/114 | 3/255
Lethargy (Nervous system disorders) | 0/228 | 0/114 | 3/255
Cerebral haemorrhage (Nervous system disorders) | 0/228 | 0/114 | 1/255
Coma (Nervous system disorders) | 0/228 | 0/114 | 1/255
Convulsion (Nervous system disorders) | 0/228 | 0/114 | 1/255
Dizziness (Nervous system disorders) | 0/228 | 0/114 | 1/255
Guillain-Barre syndrome (Nervous system disorders) | 0/228 | 0/114 | 1/255
Intracranial venous sinus thrombosis (Nervous system disorders) | 0/228 | 0/114 | 1/255
Lacunar infarction (Nervous system disorders) | 0/228 | 0/114 | 1/255
Loss of consciousness (Nervous system disorders) | 0/228 | 0/114 | 1/255
Paraesthesia (Nervous system disorders) | 0/228 | 0/114 | 1/255
Confusional state (Psychiatric disorders) | 0/228 | 0/114 | 4/255
Agitation (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Completed suicide (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Renal failure (Renal and urinary disorders) | 0/228 | 0/114 | 2/255
Renal impairment (Renal and urinary disorders) | 0/228 | 0/114 | 2/255
Dysuria (Renal and urinary disorders) | 0/228 | 0/114 | 1/255
Uterine polyp (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 3/255
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 2/255
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 2/255
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Hepatic embolisation (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Stent placement (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Hypertension (Vascular disorders) | 0/228 | 0/114 | 4/255
Hypotension (Vascular disorders) | 0/228 | 0/114 | 3/255
Thrombophlebitis (Vascular disorders) | 0/228 | 0/114 | 2/255
Embolism (Vascular disorders) | 0/228 | 0/114 | 1/255
Jugular vein thrombosis (Vascular disorders) | 0/228 | 0/114 | 1/255
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sunitinib Double-Blind Treatment | Placebo Double-Blind Treatment | Sunitinib Open-Label Treatment
Anaemia (Blood and lymphatic system disorders) | 46/228 | 10/114 | 80/255
Neutropenia (Blood and lymphatic system disorders) | 33/228 | 1/114 | 64/255
Thrombocytopenia (Blood and lymphatic system disorders) | 33/228 | 1/114 | 44/255
Leukopenia (Blood and lymphatic system disorders) | 11/228 | 1/114 | 22/255
Lymphopenia (Blood and lymphatic system disorders) | 2/228 | 1/114 | 9/255
Febrile neutropenia (Blood and lymphatic system disorders) | 1/228 | 0/114 | 2/255
Hand and foot syndrome secondary to sickle cell anaemia (Blood and lymphatic system disorders) | 1/228 | 0/114 | 0/255
Lymphadenopathy (Blood and lymphatic system disorders) | 1/228 | 0/114 | 1/255
Pancytopenia (Blood and lymphatic system disorders) | 1/228 | 0/114 | 1/255
Ejection fraction decreased (Cardiac disorders) | 19/228 | 3/114 | 5/255
Left ventricular dysfunction (Cardiac disorders) | 4/228 | 1/114 | 6/255
Tachycardia (Cardiac disorders) | 3/228 | 0/114 | 4/255
Bradycardia (Cardiac disorders) | 2/228 | 0/114 | 3/255
Cardiac disorder (Cardiac disorders) | 2/228 | 0/114 | 0/255
Cardiomyopathy (Cardiac disorders) | 2/228 | 0/114 | 1/255
Palpitations (Cardiac disorders) | 2/228 | 2/114 | 2/255
Angina pectoris (Cardiac disorders) | 1/228 | 0/114 | 3/255
Arrhythmia supraventricular (Cardiac disorders) | 1/228 | 0/114 | 0/255
Atrial fibrillation (Cardiac disorders) | 1/228 | 1/114 | 1/255
Cardiac arrest (Cardiac disorders) | 1/228 | 1/114 | 0/255
Cardiac failure (Cardiac disorders) | 1/228 | 1/114 | 1/255
Cardiomegaly (Cardiac disorders) | 1/228 | 0/114 | 0/255
Electrocardiogram QT prolonged (Cardiac disorders) | 1/228 | 0/114 | 0/255
Left atrial dilatation (Cardiac disorders) | 1/228 | 1/114 | 1/255
Left ventricular failure (Cardiac disorders) | 1/228 | 0/114 | 0/255
Mitral valve incompetence (Cardiac disorders) | 1/228 | 0/114 | 0/255
Pericardial effusion (Cardiac disorders) | 1/228 | 0/114 | 1/255
Sinus arrhythmia (Cardiac disorders) | 1/228 | 0/114 | 0/255
Ventricular extrasystoles (Cardiac disorders) | 1/228 | 0/114 | 0/255
Bundle branch block left (Cardiac disorders) | 0/228 | 1/114 | 0/255
Sinus tachycardia (Cardiac disorders) | 0/228 | 1/114 | 0/255
Pyloric stenosis (Congenital, familial and genetic disorders) | 1/228 | 0/114 | 0/255
Ear discomfort (Ear and labyrinth disorders) | 1/228 | 0/114 | 2/255
Ear pain (Ear and labyrinth disorders) | 1/228 | 1/114 | 3/255
Hypoacusis (Ear and labyrinth disorders) | 1/228 | 0/114 | 1/255
Vertigo (Ear and labyrinth disorders) | 1/228 | 1/114 | 1/255
Tinnitus (Ear and labyrinth disorders) | 0/228 | 1/114 | 3/255
Hypothyroidism (Endocrine disorders) | 9/228 | 1/114 | 45/255
Adrenal insufficiency (Endocrine disorders) | 1/228 | 0/114 | 1/255
Cushingoid (Endocrine disorders) | 1/228 | 0/114 | 0/255
Eye oedema (Eye disorders) | 5/228 | 0/114 | 5/255
Lacrimation increased (Eye disorders) | 4/228 | 1/114 | 2/255
Vision blurred (Eye disorders) | 3/228 | 1/114 | 5/255
Conjunctival haemorrhage (Eye disorders) | 2/228 | 0/114 | 0/255
Conjunctivitis (Eye disorders) | 2/228 | 2/114 | 6/255
Visual disturbance (Eye disorders) | 2/228 | 0/114 | 4/255
Diplopia (Eye disorders) | 1/228 | 2/114 | 0/255
Eyelid oedema (Eye disorders) | 1/228 | 0/114 | 9/255
Lacrimal disorder (Eye disorders) | 1/228 | 0/114 | 0/255
Photopsia (Eye disorders) | 1/228 | 0/114 | 0/255
Vitreous floaters (Eye disorders) | 1/228 | 0/114 | 1/255
Diarrhoea (Gastrointestinal disorders) | 102/228 | 21/114 | 119/255
Abdominal pain (Gastrointestinal disorders) | 82/228 | 37/114 | 106/255
Nausea (Gastrointestinal disorders) | 80/228 | 28/114 | 114/255
Vomiting (Gastrointestinal disorders) | 63/228 | 23/114 | 93/255
Constipation (Gastrointestinal disorders) | 53/228 | 22/114 | 75/255
Dyspepsia (Gastrointestinal disorders) | 45/228 | 6/114 | 56/255
Stomatitis (Gastrointestinal disorders) | 37/228 | 1/114 | 44/255
Abdominal pain upper (Gastrointestinal disorders) | 28/228 | 10/114 | 37/255
Dry mouth (Gastrointestinal disorders) | 26/228 | 4/114 | 22/255
Flatulence (Gastrointestinal disorders) | 24/228 | 5/114 | 26/255
Abdominal distension (Gastrointestinal disorders) | 18/228 | 9/114 | 38/255
Oral pain (Gastrointestinal disorders) | 16/228 | 1/114 | 30/255
Glossodynia (Gastrointestinal disorders) | 13/228 | 0/114 | 20/255
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10/228 | 2/114 | 23/255
Ascites (Gastrointestinal disorders) | 9/228 | 6/114 | 9/255
Abdominal discomfort (Gastrointestinal disorders) | 8/228 | 0/114 | 10/255
Rectal haemorrhage (Gastrointestinal disorders) | 8/228 | 2/114 | 16/255
Mouth ulceration (Gastrointestinal disorders) | 7/228 | 0/114 | 5/255
Dysphagia (Gastrointestinal disorders) | 6/228 | 1/114 | 12/255
Gastritis (Gastrointestinal disorders) | 4/228 | 0/114 | 3/255
Gingival pain (Gastrointestinal disorders) | 4/228 | 1/114 | 3/255
Haemorrhoids (Gastrointestinal disorders) | 4/228 | 2/114 | 12/255
Oral discomfort (Gastrointestinal disorders) | 4/228 | 1/114 | 3/255
Abdominal pain lower (Gastrointestinal disorders) | 3/228 | 2/114 | 8/255
Eructation (Gastrointestinal disorders) | 3/228 | 2/114 | 5/255
Lip dry (Gastrointestinal disorders) | 3/228 | 0/114 | 2/255
Oesophagitis (Gastrointestinal disorders) | 3/228 | 1/114 | 6/255
Oral mucosal discolouration (Gastrointestinal disorders) | 3/228 | 0/114 | 0/255
Proctalgia (Gastrointestinal disorders) | 3/228 | 0/114 | 7/255
Reflux oesophagitis (Gastrointestinal disorders) | 3/228 | 0/114 | 1/255
Retching (Gastrointestinal disorders) | 3/228 | 0/114 | 2/255
Salivary hypersecretion (Gastrointestinal disorders) | 3/228 | 0/114 | 0/255
Toothache (Gastrointestinal disorders) | 3/228 | 2/114 | 5/255
Duodenogastric reflux (Gastrointestinal disorders) | 2/228 | 1/114 | 2/255
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2/228 | 5/114 | 5/255
Gingival bleeding (Gastrointestinal disorders) | 2/228 | 0/114 | 1/255
Glossitis (Gastrointestinal disorders) | 2/228 | 0/114 | 6/255
Haematochezia (Gastrointestinal disorders) | 2/228 | 2/114 | 4/255
Intestinal obstruction (Gastrointestinal disorders) | 2/228 | 1/114 | 2/255
Lip pain (Gastrointestinal disorders) | 2/228 | 0/114 | 1/255
Lip ulceration (Gastrointestinal disorders) | 2/228 | 0/114 | 0/255
Melaena (Gastrointestinal disorders) | 2/228 | 1/114 | 4/255
Painful defaecation (Gastrointestinal disorders) | 2/228 | 0/114 | 2/255
Paraesthesia oral (Gastrointestinal disorders) | 2/228 | 0/114 | 1/255
Small intestinal obstruction (Gastrointestinal disorders) | 2/228 | 0/114 | 3/255
Stomach discomfort (Gastrointestinal disorders) | 2/228 | 0/114 | 4/255
Tongue blistering (Gastrointestinal disorders) | 2/228 | 0/114 | 0/255
Aerophagia (Gastrointestinal disorders) | 1/228 | 1/114 | 1/255
Anal fissure (Gastrointestinal disorders) | 1/228 | 0/114 | 1/255
Anal fistula (Gastrointestinal disorders) | 1/228 | 0/114 | 2/255
Anal inflammation (Gastrointestinal disorders) | 1/228 | 0/114 | 1/255
Anorectal discomfort (Gastrointestinal disorders) | 1/228 | 0/114 | 4/255
Aphthous stomatitis (Gastrointestinal disorders) | 1/228 | 0/114 | 1/255
Breath odour (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Chapped lips (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Cheilosis (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Colitis ulcerative (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Epigastric discomfort (Gastrointestinal disorders) | 1/228 | 0/114 | 2/255
Faecal incontinence (Gastrointestinal disorders) | 1/228 | 1/114 | 1/255
Gastric haemorrhage (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Gastric ulcer (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Gastritis haemorrhagic (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Gastrointestinal obstruction (Gastrointestinal disorders) | 1/228 | 1/114 | 1/255
Gastrointestinal pain (Gastrointestinal disorders) | 1/228 | 0/114 | 1/255
Gingival swelling (Gastrointestinal disorders) | 1/228 | 0/114 | 1/255
Haematemesis (Gastrointestinal disorders) | 1/228 | 2/114 | 6/255
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Inguinal hernia (Gastrointestinal disorders) | 1/228 | 0/114 | 2/255
Intestinal haemorrhage (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Lip swelling (Gastrointestinal disorders) | 1/228 | 0/114 | 3/255
Loose tooth (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Mouth haemorrhage (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Odynophagia (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Oesophageal haemorrhage (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Oesophageal pain (Gastrointestinal disorders) | 1/228 | 0/114 | 1/255
Oesophageal ulcer (Gastrointestinal disorders) | 1/228 | 0/114 | 2/255
Periodontal disease (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Periodontitis (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Proctitis (Gastrointestinal disorders) | 1/228 | 0/114 | 3/255
Rectal lesion (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Steatorrhoea (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Tooth discolouration (Gastrointestinal disorders) | 1/228 | 0/114 | 0/255
Enterovesical fistula (Gastrointestinal disorders) | 0/228 | 1/114 | 1/255
Faeces discoloured (Gastrointestinal disorders) | 0/228 | 1/114 | 0/255
Ileus (Gastrointestinal disorders) | 0/228 | 2/114 | 2/255
Pancreatitis acute (Gastrointestinal disorders) | 0/228 | 1/114 | 0/255
Subileus (Gastrointestinal disorders) | 0/228 | 1/114 | 1/255
Varices oesophageal (Gastrointestinal disorders) | 0/228 | 1/114 | 1/255
Fatigue (General disorders) | 104/228 | 40/114 | 156/255
Asthenia (General disorders) | 51/228 | 11/114 | 62/255
Mucosal inflammation (General disorders) | 39/228 | 0/114 | 49/255
Pyrexia (General disorders) | 39/228 | 11/114 | 52/255
Oedema peripheral (General disorders) | 30/228 | 15/114 | 73/255
Oedema (General disorders) | 17/228 | 0/114 | 14/255
Chest pain (General disorders) | 10/228 | 5/114 | 17/255
Chills (General disorders) | 8/228 | 2/114 | 9/255
Disease progression (General disorders) | 8/228 | 4/114 | 33/255
Pain (General disorders) | 8/228 | 2/114 | 13/255
Face oedema (General disorders) | 3/228 | 0/114 | 9/255
Localised oedema (General disorders) | 3/228 | 0/114 | 4/255
Early satiety (General disorders) | 2/228 | 3/114 | 9/255
Influenza like illness (General disorders) | 2/228 | 2/114 | 5/255
Malaise (General disorders) | 2/228 | 0/114 | 6/255
Chest discomfort (General disorders) | 1/228 | 0/114 | 2/255
Discomfort (General disorders) | 1/228 | 0/114 | 0/255
Drug interaction (General disorders) | 1/228 | 0/114 | 0/255
Facial pain (General disorders) | 1/228 | 0/114 | 1/255
Gait disturbance (General disorders) | 1/228 | 0/114 | 3/255
General physical health deterioration (General disorders) | 1/228 | 3/114 | 5/255
Infusion site reaction (General disorders) | 1/228 | 0/114 | 0/255
Multi-organ failure (General disorders) | 1/228 | 0/114 | 1/255
Performance status decreased (General disorders) | 1/228 | 0/114 | 2/255
Hepatic pain (Hepatobiliary disorders) | 3/228 | 1/114 | 6/255
Hyperbilirubinaemia (Hepatobiliary disorders) | 3/228 | 0/114 | 4/255
Jaundice (Hepatobiliary disorders) | 3/228 | 0/114 | 3/255
Hepatomegaly (Hepatobiliary disorders) | 2/228 | 2/114 | 2/255
Acute hepatic failure (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Bile duct stone (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Cholangitis (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Cholecystitis acute (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Cholelithiasis (Hepatobiliary disorders) | 1/228 | 0/114 | 1/255
Cholestasis (Hepatobiliary disorders) | 1/228 | 0/114 | 1/255
Hepatic failure (Hepatobiliary disorders) | 1/228 | 0/114 | 2/255
Hepatic function abnormal (Hepatobiliary disorders) | 1/228 | 0/114 | 1/255
Hepatic haemorrhage (Hepatobiliary disorders) | 1/228 | 0/114 | 1/255
Portal hypertension (Hepatobiliary disorders) | 1/228 | 0/114 | 0/255
Hypersensitivity (Immune system disorders) | 0/228 | 1/114 | 0/255
Urinary tract infection (Infections and infestations) | 10/228 | 3/114 | 22/255
Influenza (Infections and infestations) | 8/228 | 2/114 | 13/255
Upper respiratory tract infection (Infections and infestations) | 6/228 | 1/114 | 18/255
Cystitis (Infections and infestations) | 5/228 | 2/114 | 3/255
Infection (Infections and infestations) | 4/228 | 0/114 | 6/255
Nasopharyngitis (Infections and infestations) | 4/228 | 3/114 | 11/255
Oral herpes (Infections and infestations) | 4/228 | 1/114 | 4/255
Sinusitis (Infections and infestations) | 4/228 | 1/114 | 8/255
Bronchitis (Infections and infestations) | 3/228 | 1/114 | 2/255
Tooth abscess (Infections and infestations) | 3/228 | 0/114 | 1/255
Tooth infection (Infections and infestations) | 3/228 | 1/114 | 4/255
Central line infection (Infections and infestations) | 2/228 | 0/114 | 0/255
Folliculitis (Infections and infestations) | 2/228 | 0/114 | 5/255
Gastroenteritis (Infections and infestations) | 2/228 | 1/114 | 11/255
Nail infection (Infections and infestations) | 2/228 | 0/114 | 1/255
Abscess limb (Infections and infestations) | 1/228 | 0/114 | 0/255
Bacteraemia (Infections and infestations) | 1/228 | 1/114 | 2/255
Catheter sepsis (Infections and infestations) | 1/228 | 0/114 | 0/255
Furuncle (Infections and infestations) | 1/228 | 0/114 | 1/255
Gastroenteritis viral (Infections and infestations) | 1/228 | 0/114 | 1/255
Gingival abscess (Infections and infestations) | 1/228 | 0/114 | 0/255
Gingival infection (Infections and infestations) | 1/228 | 0/114 | 1/255
Herpes zoster (Infections and infestations) | 1/228 | 0/114 | 5/255
Lobar pneumonia (Infections and infestations) | 1/228 | 0/114 | 0/255
Localised infection (Infections and infestations) | 1/228 | 0/114 | 0/255
Lower respiratory tract infection (Infections and infestations) | 1/228 | 1/114 | 6/255
Mediastinitis (Infections and infestations) | 1/228 | 0/114 | 0/255
Nipple infection (Infections and infestations) | 1/228 | 0/114 | 0/255
Oral candidiasis (Infections and infestations) | 1/228 | 3/114 | 3/255
Oral fungal infection (Infections and infestations) | 1/228 | 0/114 | 0/255
Oral infection (Infections and infestations) | 1/228 | 0/114 | 0/255
Pilonidal cyst (Infections and infestations) | 1/228 | 0/114 | 0/255
Pneumonia (Infections and infestations) | 1/228 | 1/114 | 5/255
Sinusitis bacterial (Infections and infestations) | 1/228 | 0/114 | 0/255
Skin infection (Infections and infestations) | 1/228 | 0/114 | 1/255
Staphylococcal infection (Infections and infestations) | 1/228 | 0/114 | 0/255
Staphylococcal sepsis (Infections and infestations) | 1/228 | 0/114 | 0/255
Subcutaneous abscess (Infections and infestations) | 1/228 | 0/114 | 1/255
Tinea infection (Infections and infestations) | 1/228 | 0/114 | 1/255
Tinea pedis (Infections and infestations) | 1/228 | 0/114 | 3/255
Tonsillitis (Infections and infestations) | 1/228 | 0/114 | 0/255
Viral infection (Infections and infestations) | 1/228 | 1/114 | 0/255
Viral oesophagitis (Infections and infestations) | 1/228 | 0/114 | 0/255
Wound infection (Infections and infestations) | 1/228 | 0/114 | 0/255
Arthritis infective (Infections and infestations) | 0/228 | 1/114 | 0/255
Laryngitis (Infections and infestations) | 0/228 | 1/114 | 2/255
Postoperative wound infection (Infections and infestations) | 0/228 | 1/114 | 2/255
Contusion (Injury, poisoning and procedural complications) | 9/228 | 1/114 | 9/255
Procedural pain (Injury, poisoning and procedural complications) | 3/228 | 1/114 | 2/255
Back injury (Injury, poisoning and procedural complications) | 1/228 | 1/114 | 2/255
Excoriation (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 2/255
Medical device pain (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 0/255
Periorbital haematoma (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 0/255
Procedural site reaction (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 0/255
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 0/255
Spinal compression fracture (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 1/255
Spinal fracture (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 0/255
Sunburn (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 1/255
Wound dehiscence (Injury, poisoning and procedural complications) | 1/228 | 0/114 | 0/255
Fall (Injury, poisoning and procedural complications) | 0/228 | 1/114 | 3/255
Hepatic haematoma (Injury, poisoning and procedural complications) | 0/228 | 1/114 | 1/255
Injury (Injury, poisoning and procedural complications) | 0/228 | 1/114 | 1/255
Overdose (Injury, poisoning and procedural complications) | 0/228 | 1/114 | 0/255
Weight decreased (Investigations) | 14/228 | 6/114 | 45/255
Platelet count decreased (Investigations) | 9/228 | 0/114 | 13/255
Blood creatinine increased (Investigations) | 7/228 | 1/114 | 20/255
Haemoglobin decreased (Investigations) | 7/228 | 1/114 | 11/255
Lipase increased (Investigations) | 6/228 | 3/114 | 8/255
Blood amylase increased (Investigations) | 5/228 | 2/114 | 6/255
Blood bilirubin increased (Investigations) | 5/228 | 2/114 | 3/255
White blood cell count decreased (Investigations) | 5/228 | 0/114 | 12/255
Blood alkaline phosphatase increased (Investigations) | 4/228 | 2/114 | 10/255
Blood creatine phosphokinase increased (Investigations) | 4/228 | 1/114 | 2/255
Alanine aminotransferase increased (Investigations) | 3/228 | 3/114 | 8/255
Aspartate aminotransferase increased (Investigations) | 3/228 | 1/114 | 9/255
Neutrophil count decreased (Investigations) | 3/228 | 0/114 | 11/255
Urine output decreased (Investigations) | 3/228 | 1/114 | 1/255
Activated partial thromboplastin time prolonged (Investigations) | 2/228 | 0/114 | 2/255
International normalised ratio increased (Investigations) | 2/228 | 0/114 | 2/255
Prothrombin time prolonged (Investigations) | 2/228 | 0/114 | 2/255
Alanine aminotransferase abnormal (Investigations) | 1/228 | 0/114 | 0/255
Ammonia increased (Investigations) | 1/228 | 0/114 | 3/255
Aspartate aminotransferase abnormal (Investigations) | 1/228 | 0/114 | 0/255
Blood alkaline phosphatase abnormal (Investigations) | 1/228 | 0/114 | 0/255
Blood bicarbonate decreased (Investigations) | 1/228 | 2/114 | 2/255
Blood bilirubin (Investigations) | 1/228 | 0/114 | 0/255
Blood creatine phosphokinase (Investigations) | 1/228 | 1/114 | 3/255
Blood creatinine (Investigations) | 1/228 | 1/114 | 1/255
Blood magnesium decreased (Investigations) | 1/228 | 0/114 | 2/255
Blood potassium increased (Investigations) | 1/228 | 0/114 | 1/255
Blood pressure increased (Investigations) | 1/228 | 0/114 | 1/255
Blood thyroid stimulating hormone increased (Investigations) | 1/228 | 0/114 | 1/255
Blood urea increased (Investigations) | 1/228 | 1/114 | 3/255
Blood urine present (Investigations) | 1/228 | 0/114 | 0/255
Haemoglobin (Investigations) | 1/228 | 0/114 | 2/255
Heart rate increased (Investigations) | 1/228 | 0/114 | 1/255
Neutrophil count (Investigations) | 1/228 | 0/114 | 1/255
Neutrophil count normal (Investigations) | 1/228 | 1/114 | 0/255
Oxygen saturation decreased (Investigations) | 1/228 | 0/114 | 0/255
Transaminases increased (Investigations) | 1/228 | 0/114 | 3/255
Blood glucose increased (Investigations) | 0/228 | 1/114 | 3/255
Blood sodium increased (Investigations) | 0/228 | 1/114 | 0/255
Breath sounds abnormal (Investigations) | 0/228 | 1/114 | 1/255
Cardiac murmur (Investigations) | 0/228 | 1/114 | 0/255
Electrocardiogram abnormal (Investigations) | 0/228 | 1/114 | 0/255
Heart rate irregular (Investigations) | 0/228 | 1/114 | 1/255
Occult blood positive (Investigations) | 0/228 | 1/114 | 0/255
Pancreatic enzymes increased (Investigations) | 0/228 | 2/114 | 1/255
Platelet count increased (Investigations) | 0/228 | 1/114 | 2/255
Anorexia (Metabolism and nutrition disorders) | 76/228 | 19/114 | 92/255
Decreased appetite (Metabolism and nutrition disorders) | 10/228 | 5/114 | 25/255
Hypokalaemia (Metabolism and nutrition disorders) | 10/228 | 1/114 | 13/255
Dehydration (Metabolism and nutrition disorders) | 9/228 | 0/114 | 19/255
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6/228 | 1/114 | 11/255
Hyperglycaemia (Metabolism and nutrition disorders) | 4/228 | 0/114 | 10/255
Hypocalcaemia (Metabolism and nutrition disorders) | 4/228 | 1/114 | 4/255
Hypoglycaemia (Metabolism and nutrition disorders) | 4/228 | 1/114 | 6/255
Hyponatraemia (Metabolism and nutrition disorders) | 3/228 | 2/114 | 4/255
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2/228 | 0/114 | 4/255
Hyperuricaemia (Metabolism and nutrition disorders) | 2/228 | 1/114 | 3/255
Food intolerance (Metabolism and nutrition disorders) | 1/228 | 0/114 | 0/255
Hypercalcaemia (Metabolism and nutrition disorders) | 1/228 | 2/114 | 2/255
Hyperkalaemia (Metabolism and nutrition disorders) | 1/228 | 1/114 | 1/255
Hyperphosphataemia (Metabolism and nutrition disorders) | 1/228 | 1/114 | 1/255
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1/228 | 0/114 | 4/255
Hypophosphataemia (Metabolism and nutrition disorders) | 1/228 | 0/114 | 4/255
Hypoproteinaemia (Metabolism and nutrition disorders) | 1/228 | 0/114 | 0/255
Metabolic acidosis (Metabolism and nutrition disorders) | 1/228 | 0/114 | 2/255
Acidosis (Metabolism and nutrition disorders) | 0/228 | 1/114 | 0/255
Appetite disorder (Metabolism and nutrition disorders) | 0/228 | 1/114 | 0/255
Gout (Metabolism and nutrition disorders) | 0/228 | 1/114 | 2/255
Increased appetite (Metabolism and nutrition disorders) | 0/228 | 2/114 | 1/255
Malnutrition (Metabolism and nutrition disorders) | 0/228 | 1/114 | 1/255
Back pain (Musculoskeletal and connective tissue disorders) | 31/228 | 14/114 | 51/255
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28/228 | 4/114 | 46/255
Arthralgia (Musculoskeletal and connective tissue disorders) | 23/228 | 8/114 | 51/255
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15/228 | 5/114 | 27/255
Myalgia (Musculoskeletal and connective tissue disorders) | 15/228 | 4/114 | 25/255
Flank pain (Musculoskeletal and connective tissue disorders) | 9/228 | 0/114 | 10/255
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9/228 | 5/114 | 28/255
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7/228 | 1/114 | 11/255
Neck pain (Musculoskeletal and connective tissue disorders) | 6/228 | 2/114 | 12/255
Bone pain (Musculoskeletal and connective tissue disorders) | 5/228 | 2/114 | 9/255
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4/228 | 0/114 | 3/255
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2/228 | 0/114 | 4/255
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2/228 | 0/114 | 4/255
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2/228 | 3/114 | 5/255
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2/228 | 0/114 | 0/255
Exostosis (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 0/255
Fistula (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 1/255
Groin pain (Musculoskeletal and connective tissue disorders) | 1/228 | 3/114 | 5/255
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 1/255
Joint effusion (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 0/255
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 1/255
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 1/255
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 2/255
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1/228 | 0/114 | 2/255
Tendonitis (Musculoskeletal and connective tissue disorders) | 1/228 | 1/114 | 2/255
Costochondritis (Musculoskeletal and connective tissue disorders) | 0/228 | 1/114 | 0/255
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/228 | 1/114 | 1/255
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0/228 | 1/114 | 0/255
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0/228 | 1/114 | 1/255
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/228 | 0/114 | 3/255
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 1/255
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 1/255
Haemorrhagic tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 6/255
Vascular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/228 | 0/114 | 0/255
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 1/114 | 0/255
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 1/114 | 1/255
Dysgeusia (Nervous system disorders) | 54/228 | 3/114 | 57/255
Headache (Nervous system disorders) | 48/228 | 18/114 | 67/255
Dizziness (Nervous system disorders) | 22/228 | 7/114 | 31/255
Paraesthesia (Nervous system disorders) | 11/228 | 1/114 | 16/255
Hypoaesthesia (Nervous system disorders) | 8/228 | 4/114 | 12/255
Neuropathy peripheral (Nervous system disorders) | 7/228 | 2/114 | 8/255
Ageusia (Nervous system disorders) | 6/228 | 0/114 | 5/255
Peripheral sensory neuropathy (Nervous system disorders) | 5/228 | 2/114 | 5/255
Sciatica (Nervous system disorders) | 4/228 | 0/114 | 3/255
Somnolence (Nervous system disorders) | 4/228 | 2/114 | 9/255
Balance disorder (Nervous system disorders) | 3/228 | 1/114 | 0/255
Hyperaesthesia (Nervous system disorders) | 3/228 | 1/114 | 3/255
Lethargy (Nervous system disorders) | 3/228 | 1/114 | 9/255
Syncope (Nervous system disorders) | 3/228 | 1/114 | 3/255
Tremor (Nervous system disorders) | 3/228 | 1/114 | 5/255
Dizziness postural (Nervous system disorders) | 2/228 | 0/114 | 2/255
Memory impairment (Nervous system disorders) | 2/228 | 1/114 | 4/255
Migraine (Nervous system disorders) | 2/228 | 0/114 | 3/255
Parosmia (Nervous system disorders) | 2/228 | 1/114 | 0/255
Sinus headache (Nervous system disorders) | 2/228 | 1/114 | 5/255
Amnesia (Nervous system disorders) | 1/228 | 0/114 | 1/255
Ataxia (Nervous system disorders) | 1/228 | 0/114 | 0/255
Cerebral ischaemia (Nervous system disorders) | 1/228 | 0/114 | 0/255
Depressed level of consciousness (Nervous system disorders) | 1/228 | 0/114 | 2/255
Diabetic neuropathy (Nervous system disorders) | 1/228 | 0/114 | 2/255
Disturbance in attention (Nervous system disorders) | 1/228 | 1/114 | 2/255
Encephalopathy (Nervous system disorders) | 1/228 | 0/114 | 0/255
Facial palsy (Nervous system disorders) | 1/228 | 0/114 | 0/255
Head discomfort (Nervous system disorders) | 1/228 | 0/114 | 0/255
Myoclonus (Nervous system disorders) | 1/228 | 0/114 | 1/255
Peripheral motor neuropathy (Nervous system disorders) | 1/228 | 0/114 | 1/255
Restless legs syndrome (Nervous system disorders) | 1/228 | 0/114 | 1/255
Sensory disturbance (Nervous system disorders) | 1/228 | 0/114 | 1/255
Syncope vasovagal (Nervous system disorders) | 1/228 | 0/114 | 1/255
Transient ischaemic attack (Nervous system disorders) | 1/228 | 0/114 | 1/255
Burning sensation (Nervous system disorders) | 0/228 | 1/114 | 1/255
Cerebrovascular accident (Nervous system disorders) | 0/228 | 1/114 | 1/255
Coma (Nervous system disorders) | 0/228 | 1/114 | 1/255
Hemicephalalgia (Nervous system disorders) | 0/228 | 1/114 | 1/255
Neuralgia (Nervous system disorders) | 0/228 | 1/114 | 1/255
Paralysis (Nervous system disorders) | 0/228 | 1/114 | 0/255
Insomnia (Psychiatric disorders) | 25/228 | 11/114 | 34/255
Anxiety (Psychiatric disorders) | 7/228 | 2/114 | 11/255
Depression (Psychiatric disorders) | 7/228 | 2/114 | 23/255
Agitation (Psychiatric disorders) | 2/228 | 1/114 | 7/255
Confusional state (Psychiatric disorders) | 2/228 | 2/114 | 14/255
Nervousness (Psychiatric disorders) | 1/228 | 1/114 | 2/255
Sleep disorder (Psychiatric disorders) | 1/228 | 0/114 | 0/255
Depressed mood (Psychiatric disorders) | 0/228 | 1/114 | 1/255
Chromaturia (Renal and urinary disorders) | 12/228 | 2/114 | 6/255
Dysuria (Renal and urinary disorders) | 10/228 | 1/114 | 12/255
Haematuria (Renal and urinary disorders) | 6/228 | 2/114 | 8/255
Urinary retention (Renal and urinary disorders) | 4/228 | 0/114 | 3/255
Hydronephrosis (Renal and urinary disorders) | 3/228 | 3/114 | 6/255
Pollakiuria (Renal and urinary disorders) | 3/228 | 4/114 | 11/255
Polyuria (Renal and urinary disorders) | 2/228 | 0/114 | 0/255
Proteinuria (Renal and urinary disorders) | 2/228 | 1/114 | 3/255
Bladder pain (Renal and urinary disorders) | 1/228 | 0/114 | 2/255
Choluria (Renal and urinary disorders) | 1/228 | 0/114 | 1/255
Nephrotic syndrome (Renal and urinary disorders) | 1/228 | 0/114 | 0/255
Nocturia (Renal and urinary disorders) | 1/228 | 1/114 | 2/255
Oliguria (Renal and urinary disorders) | 1/228 | 0/114 | 3/255
Renal colic (Renal and urinary disorders) | 1/228 | 0/114 | 0/255
Renal failure (Renal and urinary disorders) | 1/228 | 0/114 | 2/255
Renal failure acute (Renal and urinary disorders) | 1/228 | 1/114 | 2/255
Urine odour abnormal (Renal and urinary disorders) | 1/228 | 0/114 | 2/255
Bladder spasm (Renal and urinary disorders) | 0/228 | 1/114 | 2/255
Hydroureter (Renal and urinary disorders) | 0/228 | 1/114 | 2/255
Micturition urgency (Renal and urinary disorders) | 0/228 | 1/114 | 3/255
Ureteric obstruction (Renal and urinary disorders) | 0/228 | 1/114 | 0/255
Urethral stenosis (Renal and urinary disorders) | 0/228 | 1/114 | 2/255
Urinary incontinence (Renal and urinary disorders) | 0/228 | 1/114 | 3/255
Gynaecomastia (Reproductive system and breast disorders) | 4/228 | 0/114 | 2/255
Pelvic pain (Reproductive system and breast disorders) | 4/228 | 3/114 | 11/255
Oedema genital (Reproductive system and breast disorders) | 2/228 | 0/114 | 1/255
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Genital discomfort (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Genital pain (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Genital rash (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Menstruation delayed (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Metrorrhagia (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Nipple pain (Reproductive system and breast disorders) | 1/228 | 1/114 | 0/255
Pelvic discomfort (Reproductive system and breast disorders) | 1/228 | 1/114 | 2/255
Vaginal erythema (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/228 | 0/114 | 4/255
Vaginal pain (Reproductive system and breast disorders) | 1/228 | 0/114 | 1/255
Vulval ulceration (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1/228 | 0/114 | 0/255
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/228 | 1/114 | 1/255
Breast mass (Reproductive system and breast disorders) | 0/228 | 1/114 | 2/255
Breast pain (Reproductive system and breast disorders) | 0/228 | 1/114 | 0/255
Perineal pain (Reproductive system and breast disorders) | 0/228 | 1/114 | 1/255
Prostatitis (Reproductive system and breast disorders) | 0/228 | 1/114 | 2/255
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25/228 | 16/114 | 56/255
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22/228 | 0/114 | 27/255
Cough (Respiratory, thoracic and mediastinal disorders) | 19/228 | 14/114 | 43/255
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9/228 | 3/114 | 17/255
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4/228 | 1/114 | 6/255
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4/228 | 1/114 | 7/255
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4/228 | 3/114 | 5/255
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4/228 | 0/114 | 7/255
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3/228 | 1/114 | 3/255
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2/228 | 0/114 | 1/255
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2/228 | 2/114 | 9/255
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2/228 | 0/114 | 5/255
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2/228 | 1/114 | 4/255
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 3/255
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 1/255
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 2/255
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 6/255
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 1/255
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 1/255
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 1/255
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 1/255
Rales (Respiratory, thoracic and mediastinal disorders) | 1/228 | 1/114 | 0/255
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 1/255
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1/228 | 0/114 | 0/255
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0/228 | 1/114 | 1/255
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0/228 | 1/114 | 1/255
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0/228 | 1/114 | 0/255
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/228 | 1/114 | 4/255
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0/228 | 1/114 | 1/255
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/228 | 1/114 | 0/255
Skin discolouration (Skin and subcutaneous tissue disorders) | 64/228 | 7/114 | 77/255
Rash (Skin and subcutaneous tissue disorders) | 40/228 | 7/114 | 48/255
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 25/228 | 1/114 | 56/255
Hair colour changes (Skin and subcutaneous tissue disorders) | 19/228 | 2/114 | 50/255
Dry skin (Skin and subcutaneous tissue disorders) | 17/228 | 3/114 | 33/255
Alopecia (Skin and subcutaneous tissue disorders) | 14/228 | 1/114 | 22/255
Skin reaction (Skin and subcutaneous tissue disorders) | 13/228 | 0/114 | 22/255
Pruritus (Skin and subcutaneous tissue disorders) | 11/228 | 4/114 | 21/255
Erythema (Skin and subcutaneous tissue disorders) | 10/228 | 3/114 | 18/255
Eczema (Skin and subcutaneous tissue disorders) | 8/228 | 2/114 | 14/255
Night sweats (Skin and subcutaneous tissue disorders) | 8/228 | 3/114 | 10/255
Periorbital oedema (Skin and subcutaneous tissue disorders) | 8/228 | 0/114 | 13/255
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8/228 | 0/114 | 8/255
Dermatitis (Skin and subcutaneous tissue disorders) | 6/228 | 0/114 | 6/255
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5/228 | 3/114 | 8/255
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5/228 | 0/114 | 8/255
Blister (Skin and subcutaneous tissue disorders) | 4/228 | 0/114 | 9/255
Ecchymosis (Skin and subcutaneous tissue disorders) | 4/228 | 0/114 | 6/255
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4/228 | 0/114 | 10/255
Petechiae (Skin and subcutaneous tissue disorders) | 4/228 | 0/114 | 5/255
Skin fissures (Skin and subcutaneous tissue disorders) | 4/228 | 0/114 | 8/255
Acne (Skin and subcutaneous tissue disorders) | 3/228 | 0/114 | 4/255
Nail disorder (Skin and subcutaneous tissue disorders) | 3/228 | 0/114 | 2/255
Skin lesion (Skin and subcutaneous tissue disorders) | 3/228 | 1/114 | 9/255
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2/228 | 1/114 | 0/255
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 2/228 | 0/114 | 2/255
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 2/228 | 0/114 | 2/255
Nail discolouration (Skin and subcutaneous tissue disorders) | 2/228 | 0/114 | 1/255
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2/228 | 0/114 | 4/255
Rash erythematous (Skin and subcutaneous tissue disorders) | 2/228 | 0/114 | 2/255
Rash macular (Skin and subcutaneous tissue disorders) | 2/228 | 1/114 | 2/255
Urticaria (Skin and subcutaneous tissue disorders) | 2/228 | 1/114 | 0/255
Acrodermatitis (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 5/255
Cold sweat (Skin and subcutaneous tissue disorders) | 1/228 | 1/114 | 0/255
Dermal cyst (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 2/255
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 1/255
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 0/255
Madarosis (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 0/255
Pain of skin (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 3/255
Palmar erythema (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 2/255
Plantar erythema (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 1/255
Rash generalised (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 1/255
Skin atrophy (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 0/255
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 0/255
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 2/255
Skin toxicity (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 1/255
Skin ulcer (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 3/255
Swelling face (Skin and subcutaneous tissue disorders) | 1/228 | 0/114 | 2/255
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0/228 | 1/114 | 0/255
Onychoclasis (Skin and subcutaneous tissue disorders) | 0/228 | 1/114 | 1/255
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0/228 | 1/114 | 1/255
Skin irritation (Skin and subcutaneous tissue disorders) | 0/228 | 1/114 | 3/255
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0/228 | 1/114 | 2/255
Telangiectasia (Skin and subcutaneous tissue disorders) | 0/228 | 1/114 | 2/255
Skin lesion excision (Surgical and medical procedures) | 1/228 | 0/114 | 0/255
Pneumatic compression therapy (Surgical and medical procedures) | 0/228 | 1/114 | 1/255
Hypertension (Vascular disorders) | 40/228 | 9/114 | 71/255
Hot flush (Vascular disorders) | 9/228 | 3/114 | 7/255
Deep vein thrombosis (Vascular disorders) | 4/228 | 0/114 | 5/255
Hypotension (Vascular disorders) | 3/228 | 1/114 | 6/255
Pallor (Vascular disorders) | 3/228 | 0/114 | 1/255
Haemorrhage (Vascular disorders) | 2/228 | 1/114 | 2/255
Hypertensive crisis (Vascular disorders) | 2/228 | 0/114 | 3/255
Vasculitis (Vascular disorders) | 2/228 | 0/114 | 0/255
Venous thrombosis limb (Vascular disorders) | 2/228 | 0/114 | 0/255
Lymphoedema (Vascular disorders) | 1/228 | 0/114 | 0/255
Orthostatic hypotension (Vascular disorders) | 1/228 | 0/114 | 1/255
Systolic hypertension (Vascular disorders) | 1/228 | 0/114 | 0/255
Thrombosis (Vascular disorders) | 1/228 | 0/114 | 0/255
Vasodilatation (Vascular disorders) | 1/228 | 0/114 | 1/255
Circulatory collapse (Vascular disorders) | 0/228 | 1/114 | 0/255
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0/228 | 0/114 | 1/255
Granulocytopenia (Blood and lymphatic system disorders) | 0/228 | 0/114 | 1/255
haemolytic anaemia (Blood and lymphatic system disorders) | 0/228 | 0/114 | 1/255
Leukocytosis (Blood and lymphatic system disorders) | 0/228 | 0/114 | 1/255
Cardiac failure congestive (Cardiac disorders) | 0/228 | 0/114 | 2/255
Cardio-respiratory arrest (Cardiac disorders) | 0/228 | 0/114 | 2/255
Sinus bradycardia (Cardiac disorders) | 0/228 | 0/114 | 2/255
Ventricular hypokinesia (Cardiac disorders) | 0/228 | 0/114 | 2/255
Left ventricular hypertrophy (Cardiac disorders) | 0/228 | 0/114 | 1/255
Myocardial infarction (Cardiac disorders) | 0/228 | 0/114 | 1/255
Myocardial ischaemia (Cardiac disorders) | 0/228 | 0/114 | 1/255
Splinter haemorhages (Cardiac disorders) | 0/228 | 0/114 | 1/255
Supraventricular tachycardia (Cardiac disorders) | 0/228 | 0/114 | 1/255
Ventricular dysfunction (Cardiac disorders) | 0/228 | 0/114 | 1/255
Dermoid cyst (Congenital, familial and genetic disorders) | 0/228 | 0/114 | 1/255
Epidermolysis (Congenital, familial and genetic disorders) | 0/228 | 0/114 | 1/255
Hydrocele (Congenital, familial and genetic disorders) | 0/228 | 0/114 | 1/255
Dysacusis (Ear and labyrinth disorders) | 0/228 | 0/114 | 1/255
Hearing impaired (Ear and labyrinth disorders) | 0/228 | 0/114 | 1/255
Hyperthyroidism (Endocrine disorders) | 0/228 | 0/114 | 3/255
Thyroid disorder (Endocrine disorders) | 0/228 | 0/114 | 1/255
Eye pain (Eye disorders) | 0/228 | 0/114 | 3/255
Eye pruritus (Eye disorders) | 0/228 | 0/114 | 3/255
Dry eye (Eye disorders) | 0/228 | 0/114 | 2/255
Glaucoma (Eye disorders) | 0/228 | 0/114 | 2/255
Macular degeneration (Eye disorders) | 0/228 | 0/114 | 2/255
Orbital oedema (Eye disorders) | 0/228 | 0/114 | 2/255
Asthenopia (Eye disorders) | 0/228 | 0/114 | 1/255
Blepharitis (Eye disorders) | 0/228 | 0/114 | 1/255
Eye discharge (Eye disorders) | 0/228 | 0/114 | 1/255
Eye haemorrhage (Eye disorders) | 0/228 | 0/114 | 1/255
Eye irritation (Eye disorders) | 0/228 | 0/114 | 1/255
Eye swelling (Eye disorders) | 0/228 | 0/114 | 1/255
Ocular hyperaemia (Eye disorders) | 0/228 | 0/114 | 1/255
Punctate keratitis (Eye disorders) | 0/228 | 0/114 | 1/255
Scleral haemorrhage (Eye disorders) | 0/228 | 0/114 | 1/255
Visual acuity reduced (Eye disorders) | 0/228 | 0/114 | 1/255
Abdominal tenderness (Gastrointestinal disorders) | 0/228 | 0/114 | 3/255
Hiatus hernia (Gastrointestinal disorders) | 0/228 | 0/114 | 3/255
Anal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 2/255
Gingivitis (Gastrointestinal disorders) | 0/228 | 0/114 | 2/255
Peritoneal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 2/255
Rectal tenesmus (Gastrointestinal disorders) | 0/228 | 0/114 | 2/255
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 2/255
Abdominal hernia (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Abdominal mass (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Abdominal rigidity (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Defaecation urgency (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Dental caries (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Diverticulum (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Duodenal fistula (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Duodenal ulcer (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Enamel anomaly (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Enterocutaneous fistula (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Gastrointestinal disorder (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Hyperchlorhydria (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Hypoaesthesia oral (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Large intestinal haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Salivary gland enlargement (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Sensitivity of teeth (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Swollen tongue (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Tongue disorder (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Tongue haemorrhage (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Tongue spasm (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Tongue ulceration (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Tooth erosion (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Umbilical hernia (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Feeling hot (General disorders) | 0/228 | 0/114 | 2/255
Ill-defined disorder (General disorders) | 0/228 | 0/114 | 2/255
Impaired healing (General disorders) | 0/228 | 0/114 | 2/255
Catheter related complication (General disorders) | 0/228 | 0/114 | 1/255
Catheter site discharge (General disorders) | 0/228 | 0/114 | 1/255
Catheter site excoriation (General disorders) | 0/228 | 0/114 | 1/255
Catheter site pain (General disorders) | 0/228 | 0/114 | 1/255
Cyst (General disorders) | 0/228 | 0/114 | 1/255
Effusion (General disorders) | 0/228 | 0/114 | 1/255
Feeling cold (General disorders) | 0/228 | 0/114 | 1/255
Hernia pain (General disorders) | 0/228 | 0/114 | 1/255
Infusion site extravasation (General disorders) | 0/228 | 0/114 | 1/255
Irritability (General disorders) | 0/228 | 0/114 | 1/255
Mucosal dryness (General disorders) | 0/228 | 0/114 | 1/255
Necrosis (General disorders) | 0/228 | 0/114 | 1/255
Peripheral coldness (General disorders) | 0/228 | 0/114 | 1/255
Pneumatosis (General disorders) | 0/228 | 0/114 | 1/255
Thirst (General disorders) | 0/228 | 0/114 | 1/255
Ulcer haemorrhage (General disorders) | 0/228 | 0/114 | 1/255
Xerosis (General disorders) | 0/228 | 0/114 | 1/255
Hepatotoxicity (Hepatobiliary disorders) | 0/228 | 0/114 | 2/255
Portal vein thrombosis (Hepatobiliary disorders) | 0/228 | 0/114 | 2/255
Cholecystitis (Hepatobiliary disorders) | 0/228 | 0/114 | 1/255
Foetor hepaticus (Hepatobiliary disorders) | 0/228 | 0/114 | 1/255
Seasonal allergy (Immune system disorders) | 0/228 | 0/114 | 1/255
Respiratory tract infection (Infections and infestations) | 0/228 | 0/114 | 5/255
Rhinitis (Infections and infestations) | 0/228 | 0/114 | 6/255
Cellulitis (Infections and infestations) | 0/228 | 0/114 | 3/255
Ear infection (Infections and infestations) | 0/228 | 0/114 | 3/255
Pharyngitis (Infections and infestations) | 0/228 | 0/114 | 3/255
Sepsis (Infections and infestations) | 0/228 | 0/114 | 3/255
Abdominal abscess (Infections and infestations) | 0/228 | 0/114 | 1/255
Anal infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Bacterial infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Campylobacter infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Diverticulitis (Infections and infestations) | 0/228 | 0/114 | 1/255
Empyema (Infections and infestations) | 0/228 | 0/114 | 1/255
Fungal infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Gastrointestinal infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Genital herpes (Infections and infestations) | 0/228 | 0/114 | 1/255
Herpes simplex (Infections and infestations) | 0/228 | 0/114 | 1/255
Infected skin ulcer (Infections and infestations) | 0/228 | 0/114 | 1/255
Liver abscess (Infections and infestations) | 0/228 | 0/114 | 1/255
Lung infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Necrotising ulcerative gingivostomatitis (Infections and infestations) | 0/228 | 0/114 | 1/255
Oesophageal candidiasis (Infections and infestations) | 0/228 | 0/114 | 1/255
Orchitis (Infections and infestations) | 0/228 | 0/114 | 1/255
Osteomyelitis (Infections and infestations) | 0/228 | 0/114 | 1/255
Otitis media (Infections and infestations) | 0/228 | 0/114 | 1/255
Perirectal abscess (Infections and infestations) | 0/228 | 0/114 | 1/255
Proctitis monilial (Infections and infestations) | 0/228 | 0/114 | 1/255
Pyelonephritis (Infections and infestations) | 0/228 | 0/114 | 1/255
Urinary tract infection fungal (Infections and infestations) | 0/228 | 0/114 | 1/255
Urosepsis (Infections and infestations) | 0/228 | 0/114 | 1/255
Viral upper respiratory tract infection (Infections and infestations) | 0/228 | 0/114 | 1/255
Skin laceration (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 4/255
Thermal burn (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 2/255
Wound (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 2/255
Anal injury (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Device malfunction (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Feeding tube complication (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Joint sprain (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Ligament rupture (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Limb injury (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Medical device complication (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Medical device site reaction (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Medication error (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Muscle strain (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Neck injury (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Post gastric surgery syndrome (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Postoperative constipation (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Postoperative fever (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Skeletal injury (Injury, poisoning and procedural complications) | 0/228 | 0/114 | 1/255
Weight increased (Investigations) | 0/228 | 0/114 | 6/255
Blood lactate dehydrogenase increased (Investigations) | 0/228 | 0/114 | 5/255
Blood potassium decreased (Investigations) | 0/228 | 0/114 | 4/255
Blood uric acid increased (Investigations) | 0/228 | 0/114 | 4/255
Blood albumin decreased (Investigations) | 0/228 | 0/114 | 3/255
Liver function test abnormal (Investigations) | 0/228 | 0/114 | 2/255
Platelet count (Investigations) | 0/228 | 0/114 | 2/255
Bacterial culture positive (Investigations) | 0/228 | 0/114 | 1/255
Blood alkaline phosphatase (Investigations) | 0/228 | 0/114 | 1/255
Blood calcium decreased (Investigations) | 0/228 | 0/114 | 1/255
Blood glucose decreased (Investigations) | 0/228 | 0/114 | 1/255
Blood phosphorus decreased (Investigations) | 0/228 | 0/114 | 1/255
C-reactive protein increased (Investigations) | 0/228 | 0/114 | 1/255
ECG signs of myocardial ischaemia (Investigations) | 0/228 | 0/114 | 1/255
Electrocardiogram ST segment depression (Investigations) | 0/228 | 0/114 | 1/255
Gamma-glutamyltransferase increased (Investigations) | 0/228 | 0/114 | 1/255
Hepatic enzyme increased (Investigations) | 0/228 | 0/114 | 1/255
Lymph node palpable (Investigations) | 0/228 | 0/114 | 1/255
Lymphocyte count decreased (Investigations) | 0/228 | 0/114 | 1/255
Mean cell volume increased (Investigations) | 0/228 | 0/114 | 1/255
Multiple gated acquisition scan abnormal (Investigations) | 0/228 | 0/114 | 1/255
Venous pressure jugular increased (Investigations) | 0/228 | 0/114 | 1/255
Vitamin B12 decreased (Investigations) | 0/228 | 0/114 | 1/255
White blood cell count (Investigations) | 0/228 | 0/114 | 1/255
White blood cell count increased (Investigations) | 0/228 | 0/114 | 1/255
Hypomagnesaemia (Metabolism and nutrition disorders) | 0/228 | 0/114 | 5/255
Cachexia (Metabolism and nutrition disorders) | 0/228 | 0/114 | 2/255
Cow's milk intolerance (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Fluid retention (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Hypochloraemia (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Iron deficiency (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Lactose intolerance (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Polydipsia (Metabolism and nutrition disorders) | 0/228 | 0/114 | 1/255
Arthritis (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Joint swelling (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Myopathy (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0/228 | 0/114 | 1/255
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 3/255
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/228 | 0/114 | 1/255
Hepatic encephalopathy (Nervous system disorders) | 0/228 | 0/114 | 5/255
Dysarthria (Nervous system disorders) | 0/228 | 0/114 | 2/255
Loss of consciousness (Nervous system disorders) | 0/228 | 0/114 | 2/255
Aphonia (Nervous system disorders) | 0/228 | 0/114 | 1/255
Asterixis (Nervous system disorders) | 0/228 | 0/114 | 1/255
Carotid artery disease (Nervous system disorders) | 0/228 | 0/114 | 1/255
Cerebral haemorrhage (Nervous system disorders) | 0/228 | 0/114 | 1/255
Cervical root pain (Nervous system disorders) | 0/228 | 0/114 | 1/255
Convulsion (Nervous system disorders) | 0/228 | 0/114 | 1/255
Dysaesthesia (Nervous system disorders) | 0/228 | 0/114 | 1/255
Guillain-barre syndrome (Nervous system disorders) | 0/228 | 0/114 | 1/255
Hemiparesis (Nervous system disorders) | 0/228 | 0/114 | 1/255
Hypogeusia (Nervous system disorders) | 0/228 | 0/114 | 1/255
Intention tremor (Nervous system disorders) | 0/228 | 0/114 | 1/255
Intracranial venous sinus thrombosis (Nervous system disorders) | 0/228 | 0/114 | 1/255
Lacunar infarction (Nervous system disorders) | 0/228 | 0/114 | 1/255
Migraine with aura (Nervous system disorders) | 0/228 | 0/114 | 1/255
Movement disorder (Nervous system disorders) | 0/228 | 0/114 | 1/255
Petit mal epilepsy (Nervous system disorders) | 0/228 | 0/114 | 1/255
Mood altered (Psychiatric disorders) | 0/228 | 0/114 | 2/255
Abnormal dreams (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Apathy (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Completed suicide (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Dysphemia (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Emotional disorder (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Hallucination (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Psychomotor retardation (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Psychotic disorder (Psychiatric disorders) | 0/228 | 0/114 | 1/255
Renal impairment (Renal and urinary disorders) | 0/228 | 0/114 | 3/255
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0/228 | 0/114 | 1/255
Obstructive uropathy (Renal and urinary disorders) | 0/228 | 0/114 | 1/255
Renal cyst (Renal and urinary disorders) | 0/228 | 0/114 | 1/255
Residual urine (Renal and urinary disorders) | 0/228 | 0/114 | 1/255
Scrotal oedema (Reproductive system and breast disorders) | 0/228 | 0/114 | 3/255
Erectile dysfunction (Reproductive system and breast disorders) | 0/228 | 0/114 | 2/255
Genital haemorrhage (Reproductive system and breast disorders) | 0/228 | 0/114 | 2/255
Genital lesion (Reproductive system and breast disorders) | 0/228 | 0/114 | 2/255
Genital rash (Reproductive system and breast disorders) | 0/228 | 0/114 | 2/255
Balanoposthitis (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Breast swelling (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Dyspareunia (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Genital erythema (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Menstruation irregular (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Penile haemorrhage (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Penile oedema (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Perineal fistula (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Pruritus genital (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Uterine polyp (Reproductive system and breast disorders) | 0/228 | 0/114 | 1/255
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 2/255
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 2/255
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 2/255
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0/228 | 0/114 | 1/255
Purpura (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 5/255
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 4/255
Skin disorder (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 4/255
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 3/255
Yellow skin (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 3/255
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 2/255
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Blood blister (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Dermatosis (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Prurigo (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Psoriasis (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Skin chapped (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Skin induration (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0/228 | 0/114 | 1/255
Cyst drainage (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Debridement (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Hepatic embolisation (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Mediastinal operation (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Packed red blood cell transfusion (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Sinus operation (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Stent placement (Surgical and medical procedures) | 0/228 | 0/114 | 1/255
Flushing (Vascular disorders) | 0/228 | 0/114 | 4/255
Thrombophlebitis (Vascular disorders) | 0/228 | 0/114 | 2/255
Embolism (Vascular disorders) | 0/228 | 0/114 | 1/255
Essential hypertension (Vascular disorders) | 0/228 | 0/114 | 1/255
Jugular vein thrombosis (Vascular disorders) | 0/228 | 0/114 | 1/255
Peripheral ischaemia (Vascular disorders) | 0/228 | 0/114 | 1/255
Phlebitis (Vascular disorders) | 0/228 | 0/114 | 1/255
Cheilitis (Gastrointestinal disorders) | 0/228 | 0/114 | 3/255
Colitis (Gastrointestinal disorders) | 0/228 | 0/114 | 1/255
Blood sodium decreased (Investigations) | 0/228 | 0/114 | 2/255

LIMITATIONS AND CAVEATS:
Duration of Tumor Response could not be reliably estimated at the time of analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.